CLINICAL TRIAL: NCT06160960
Title: Influence of Pupillary Behavior During Eye Surgery on Morphological and Functional Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Klinikum Klagenfurt am Wörthersee (Other)
Collaborators: University of Klagenfurt (Other)
Responsible Party: Principal Investigator, Yosuf El-Shabrawi, Prim. Univ. Prof. Dr. Yosuf El-Shabrawi, Klinikum Klagenfurt am Wörthersee
Other Study IDs: A 28/17
Record Dates: First submitted 2023-11-25; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Cataract; Corneal Disease; Vitreous Disorder
Keywords: Cataract; refractive surgery; vitrectomy
MeSH Terms: conditions — Cataract; Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: OCT Scan, Video of pupil movement, video of toric lens — A picture of the central macular area is taken, video of pupil movment, video of toric lens rotation.

SUMMARY:
Pupillary movement during eye surgery can be a challenge for eye surgeons. Despite the risk of intraocular lens damage and malpositioning due to mechanical manipulation1, iris manipulation may lead to a significant elevation of cytokines in the aqueous humor and an increase of postoperative inflammation2, 3. Iris damage is also known to lead to an increase of prostaglandin production which will not only lead to an increase of inflammation but also has an impact on intraoperative miosis4. This leads to the assumption that postoperative inflammation can be related to intraoperative pupillary movements due to the same leading cause of an increase of inflammatory mediators. Tracking intraoperative pupillary movements might therefore be a helpful tool for the prediction of postoperative PCME and could have an impact on therapeutic decisions after surgery.

ELIGIBILITY:
Inclusion Criteria:

* presence of significant cataract,
* written consent.
* presence of other ocular conditions requiring surgery such as: degenerative corneal disease, retinal conditions (i.e. macular pucker)

Exclusion Criteria:

- reasons for poor video quality (such as poor red reflex due to abnormal anatomy)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients receiving surgery and that want to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
pupillary movement | during surgery
  Analyzing the extend of pupil movement during cataract surgery
IOL rotation | Video taken immediately postoperative and 2-4 weeks postoperative
  The rotation of the IOL directly after surgery and a 2-4 weeks postoperative when the second eye is operated.
retinal thickness | at baseline and 2-4 weeks postoperative
  OCT Scan to measure retinal thickness at baseline and 2-4 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- KlinikumKlagenfurt, Klagenfurt, Carinthia, Austria

REFERENCES:
- [Result] Singh A, Kapoor G, Baranwal VK, Kalra N. Rotational stability of Toric intraocular lenses. Med J Armed Forces India. 2022 Jan;78(1):68-73. doi: 10.1016/j.mjafi.2020.03.014. Epub 2020 Jul 9. PMID 35035046
- [Result] Aketa N, Yamaguchi T, Suzuki T, Higa K, Yagi-Yaguchi Y, Satake Y, Tsubota K, Shimazaki J. Iris Damage Is Associated With Elevated Cytokine Levels in Aqueous Humor. Invest Ophthalmol Vis Sci. 2017 May 1;58(6):BIO42-BIO51. doi: 10.1167/iovs.17-21421. PMID 28475702
- [Result] Williams ER, Patnaik JL, Miller DC, Lynch AM, Davidson RS, Kahook MY, Seibold LK. Iris manipulation during phacoemulsification: intraoperative and postoperative complications. Int J Ophthalmol. 2021 May 18;14(5):676-683. doi: 10.18240/ijo.2021.05.06. eCollection 2021. PMID 34012881
- [Result] AMBACHE N, KAVANAGH L, WHITING J. EFFECT OF MECHANICAL STIMULATION ON RABBITS' EYES: RELEASE OF ACTIVE SUBSTANCE IN ANTERIOR CHAMBER PERFUSATES. J Physiol. 1965 Feb;176(3):378-408. doi: 10.1113/jphysiol.1965.sp007557. No abstract available. PMID 14289827